CLINICAL TRIAL: NCT01530386
Title: A Multicenter, Open-label Study to Determine the Effects of Lacosamide on Sleep in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SP1031
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Subjects
Keywords: Lacosamide; Vimpat
MeSH Terms: interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): 300 mg/day
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide will be given orally in 50 mg tablets twice a day for 7 days. The dose will increase weekly by 100 mg per day to a target dose of 300 mg per day. Once the target dose of 300 mg per day has been achieved for 9 days, a 2-day tapering of Lacosamide will occur by 100 mg per day.

SUMMARY:
The effects of Lacosamide, an antiepileptic drug, on sleep have not been formally evaluated. The present study is being conducted to assess the effects of Lacosamide on sleep quality in healthy subjects.

DETAILED DESCRIPTION:
In some patients with Epilepsy, seizure activity is associated with specific phases of sleep/wake cycle, and sleep deprivation is known to precipitate seizure activity. Inadequate or disturbed sleep and excessive daytime drowsiness is often reported by patients with Epilepsy due to the effects of seizures as well as antiepileptic drugs. Thus, the use of healthy subjects improves the certainty that any changes in sleep are related to the study drug and not other factors.

ELIGIBILITY:
Inclusion Criteria:

* Reliable and capable subject who signs an IRB approved consent form
* Subject is male or female between 18 and 50 years old whose normal Body Mass Index (BMI) is between 18 and 28 kg/m^2
* Subject has no clinically relevant cardiovascular, renal, gastrointestinal, hepatic, metabolic, endocrine, neurological or psychiatric abnormalities
* Subject is in good health who has good sleep hygiene and normal bed times between 21:00 and 01:00 hours

Exclusion Criteria:

* Subjects who have participated in previous Lacosamide studies or received Lacosamide
* Subjects who have received another investigational medication within 30 days or currently participating in an investigational study
* Subject has a history of or screening polysomnography that reveals sleep disorders (i.e. sleep apnea or narcolepsy)
* Subject consumes more than 400 mg of caffeine per day
* Subject has known hypersensitivity to Lacosamide
* Subject has alcohol or drug abuse within last 2 years
* Subject who consumes more than 40 g of alcohol per day
* Subject has a positive alcohol breath test or urine drug screen
* Subject smokes more than half a pack of cigarettes per day or consumes nicotine products
* Subject is pregnant / nursing or child-bearing potential female not sterile or using contraception methods
* Subject is male who does not agree to use contraception
* Subjects taking any medications currently or within 2 weeks prior to first dose except non-steroidal anti-inflammatory drugs, oral contraceptives, and non-psychoactive supplements
* Subject has elevated live enzymes greater than 2 times the upper limit of normal
* Subject has donated blood or had blood loss greater than 400 mL within 3 months prior to first dose
* Subject has out of range hematology or chemistry parameters
* Subject has clinically relevant abnormality in physical examination or vital signs
* Subject has sick sinus syndrome without a pace maker or second or third degree atrioventricular block or clinically significant electrocardiogram finding
* Subject has sodium channelopathy
* Subject has experienced a myocardial infarction in last 3 months
* Subject has New York Heart Association Class III or IV heart failure
* Subject has a lifetime history of suicide attempts
* Subject has any medical or psychiatric condition
* Subject has a known history or severe anaphylactic reaction or serious blood dyscrasias

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change In Wake After Sleep Onset From Baseline To The End Of The Treatment Period | Baseline to end of Treatment Period (approximately 22 days)
  Wake after sleep onset is defined as the total time that is scored as awake in a polysomnography occurring between sleep onset and final wake-up.

SECONDARY OUTCOMES:
Change In Sleep Efficiency From Baseline To The End Of The Treatment Period | Baseline to end of Treatment Period (approximately 22 days)
  Sleep efficiency is the percentage calculated by taking the total sleep time divided by the time in bed.
Change In Total Sleep Time From Baseline To The End Of The Treatment Period | Baseline to end of Treatment Period (approximately 22 days)
  Total Sleep Time is the total of all sleep epochs within time in bed.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 877-822-9493
Locations (4):
- United States (4):
  - 005, Little Rock, Arkansas
  - 003, Cleveland, Ohio
  - 004, Austin, Texas
  - 001, Fredericksburg, Virginia

REFERENCES:
- [Derived] Hudson JD, Guptill JT, Byrnes W, Yates SL, Williams P, D'Cruz O. Assessment of the effects of lacosamide on sleep parameters in healthy subjects. Seizure. 2015 Feb;25:155-9. doi: 10.1016/j.seizure.2014.10.012. Epub 2014 Oct 25. PMID 25468512